CLINICAL TRIAL: NCT01907217
Title: A Randomised Controlled Trial of Standard Bilateral Electroconvulsive Therapy Versus High-dose Unilateral Electroconvulsive Therapy for Severe Depression
Brief Title: Enhancing the Effectiveness of Electroconvulsive Therapy in Severe Depression
Acronym: EFFECT-Dep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Patrick's Hospital, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof Declan McLoughlin, Professor, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRA/2007/5; ISRCTN23577151 (Registry Identifier: Current Controlled Trials)
Record Dates: First submitted 2013-06-16; First posted 2013-07-24 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: Electroconvulsive therapy; ECT; electrode placement; effectiveness; cognition; autobiographical memory
MeSH Terms: conditions — Depression | interventions — Methohexital; Succinylcholine; halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral ECT Mecta 5000M (Active Comparator): Modified bilateral ECT (bitemporal electrode positions) twice weekly at 1.5 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Interventions: Device: ECT Mecta 5000M; Drug: Methohexitone; Drug: Suxamethonium
- High-dose unilateral ECT Mecta 5000M (Experimental): High-dose right modified unilateral ECT twice weekly at 6 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Interventions: Device: ECT Mecta 5000M; Drug: Methohexitone; Drug: Suxamethonium

INTERVENTIONS:
Device: ECT Mecta 5000M — ECT is administered twice weekly with hand-held electrodes using the Mecta 5000M device following a standard stimulus dosing protocol. Seizure duration is measured by EEG monitoring. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0 mg/kg) as muscle relaxant. Seizure threshold (ST) is established by a method of limits at the first session and subsequent treatments will be given at 1.5 x ST for BT ECT and 6.0 x ST for RUL ECT. To reflect routine clinical practice, number of ECT treatments is determined by referring physicians who will be blind to randomisation. The treatment period varies between patients to allow up to 12 administrations of ECT, i.e. up to 6 weeks.
  Other Names: electroconvulsive therapy Mecta 500M device
Drug: Methohexitone — Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia along with suxamethonium (0.5-1.0 mg/kg)for muscle relaxation. Anesthesia is the same for both arms of the trial.
  Other Names: methohexital; Brevimytal (Hikma, Germany)
Drug: Suxamethonium — Suxamethonium (0.5-1.0 mg/kg)is used for muscle relaxation along with Methohexitone (0.75-1.0 mg/kg) for anaesthesia. Anesthesia is the same for both arms of the trial.
  Other Names: Succinylcholine; Anectine (GlaxoSmithKline, UK)

SUMMARY:
Electroconvulsive therapy (ECT) is the most powerful antidepressant treatment available and is often life-saving. There are concerns, however, that standard bitemporal ECT (the most commonly used form of ECT worldwide) causes persisting retrograde amnesia. However, clinical trials have indicated that high-dose unilateral ECT may be as effective as bitemporal ECT but have much less cognitive side-effects.

The trial aims to test the primary experimental hypothesis: High-dose (6 x ST) right unilateral ECT is as effective as (i.e. not inferior to) standard (1.5 x ST) bitemporal ECT for severe depression in terms of Hamilton Depression Rating Score (HDRS) at the end of the treatment course.

DETAILED DESCRIPTION:
The study is a two-group parallel design randomised controlled non-inferiority trial and has been registered (ISRCTN23577151). Consented patients with major depressive disorder (DSM-IV) will be randomly allocated to a course of bitemporal (BT) ECT (1.5 x ST) or high-dose right unilateral (RUL) ECT (6.0 x ST). To facilitate generalizability of results, the trial takes place under "real world" conditions and so both groups continue usual care and medications during the treatment phase and thereafter. Patients are followed-up for 12 months after completing their allocated course of ECT. Completion of the primary outcome depression-rating measure (i.e. HDRS) and the secondary outcome of most interest (autobiographical memory, using the AMI-SF) will be prioritised in the data collection.

Patients, their treating clinicians and raters are blind to treatment; clinicians administering ECT are not involved in post randomisation assessments or formal data analysis. Success of blinding for patients and raters will be assessed after the second and final treatments. The trial statistician is also blinded to allocation status.

Sample size: In a large series (n = 253) of depressed patients, Petrides et al. (2001) found a mean (SD) reduction in 24-item HDRS of 25.6 (9.4) after treatment with bitemporalT ECT (1.5 x ST). We therefore estimate that 69 patients will be required per treatment group to have 80% power to demonstrate, using a one-sided equivalence t-test at 5% level, that mean reduction in 24-item HDRS achieved using high-dose RUL ECT is no more than 4 points (i.e. equivalent to 3 points on 17-item HDRS) less than that achieved using standard BT ECT, assuming a common within-group SD of change scores of 9.4 and equal expected group mean change scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years diagnosed with major depressive episode (DSM-IV) and referred for ECT

Exclusion Criteria:

* Any condition rendering patients medically unfit for general anaesthesia or ECT; treatment with ECT in previous six months; dementia or other Axis 1 diagnosis; alcohol/other substance abuse in previous six months; inability/refusal to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-05; Primary Completion 2013-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Declan M McLoughlin, PhD, Principal Investigator — St Patrick's University Hospital
Locations (1):
- St Patrick's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
We are continuing to analyze trial data for secondary analyses. Requests for IPD will be considered where appropriate.

REFERENCES:
- [Derived] Fenton C, McLoughlin DM. Usefulness of Hamilton rating scale for depression subset scales and full versions for electroconvulsive therapy. PLoS One. 2021 Nov 9;16(11):e0259861. doi: 10.1371/journal.pone.0259861. eCollection 2021. PMID 34752484

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral ECT Mecta 5000M: Twice-weekly modified bilateral ECT (bitemporal electrode positions) twice weekly at 1.5 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Seizure threshold (ST) is established by a method of limits at the first session and subsequent treatments will be given at 1.5 x ST for BT ECT and 6.0 x ST for RUL ECT. To reflect routine clinical practice, number of ECT treatments is determined by referring physicians who will be blind to randomisation. The treatment period varies between patients to allow up to 12 administrations of ECT, i.e. up to 6 weeks.
- High-dose Unilateral ECT Mecta 5000M: Twice-weekly high-dose right modified unilateral ECT twice weekly at 6 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Seizure threshold (ST) is established by a method of limits at the first session and subsequent treatments will be given at 6.0 x ST for RUL ECT. To reflect routine clinical practice, number of ECT treatments is determined by referring physicians who will be blind to randomisation. The treatment period varies between patients to allow up to 12 administrations of ECT, i.e. up to 6 weeks.
Period: Overall Study
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Started | 69 | 69
Completed | 69 | 67
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.4) | 56.6 (15.3) | 56.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 87
  Male | 22 | 29 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 69 | 69 | 138
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS)
Description: The HDRS was originally designed to assess severity of depressive symptoms in patients with a primary depressive illness and is now the most commonly used measure of depression severity. It was first published in a 17-item format with the optional addition of 4 items making up the 21-item version. In addition to the original 21 items, the 24-item HDRS includes items on helplessness, hopelessness and worthlessness; its score range is 0-77, with higher scores reflecting greater burden of depressive symptoms.
Time Frame: HDRS scores were obtained at baseline, end of allocated ECT treatment, and at 3 and 6 month follow-up timepoints.
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bilateral ECT Mecta 5000M: Modified bilateral ECT (bitemporal electrode positions) twice weekly at 1.5 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Seizure duration is measured by EEG monitoring. Seizure threshold (ST) is established by a method of limits at the first session and subsequent treatments will be given at 1.5 x ST for BT ECT and 6.0 x ST for RUL ECT. To reflect routine clinical practice, number of ECT treatments is determined by referring physicians who will be blind to randomisation. The treatment period varies between patients to allow up to 12 administrations of ECT, i.e. up to 6 weeks.
- High-dose Unilateral ECT Mecta 5000M: Modified high-dose right modified unilateral ECT twice weekly at 6 times the seizure threshold. Methohexitone (0.75-1.0 mg/kg) is used for anaesthesia with suxamethonium (0.5-1.0mg/kg) for muscle relaxation.
  Seizure threshold (ST) is established by a method of limits at the first session and subsequent treatments will be given at 1.5 x ST for BT ECT and 6.0 x ST for RUL ECT. To reflect routine clinical practice, number of ECT treatments is determined by referring physicians who will be blind to randomisation. The treatment period varies between patients to allow up to 12 administrations of ECT, i.e. up to 6 weeks.
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Number analyzed (Participants) | 69 | 69
units on a scale
  Baseline | 29.5 (6.3) | 30.4 (6.1)
  End-of-treatment: number analyzed (Participants) | 69 | 67
  End-of-treatment | 12.5 (9.2) | 11.1 (7.5)
  3 months follow-up: number analyzed (Participants) | 53 | 60
  3 months follow-up | 15.0 (10.2) | 11.5 (9.1)
  6 months follow-up: number analyzed (Participants) | 50 | 55
  6 months follow-up | 13.0 (8.6) | 12.6 (10.9)
Statistical Analysis 1: Comparison: Bilateral ECT Mecta 5000M vs High-dose Unilateral ECT Mecta 5000M; Based on a large bitemporal ECT series, we estimated that 69 patients were required per group to have 80% power to demonstrate, using a one-sided equivalence t test at 5% level, that the mean reduction in the 24-item HAM-D score following high-dose unilateral ECT was no more than 4 points (i.e., equivalent to 3 points on the 17-item HAM-D, deemed to be clinically relevant [30]) less than that achieved using bitemporal ECT; Test type: Non-Inferiority or Equivalence — The prespecified noninferiority margin was no more than a -4 point difference at the end of treatment between the bilateral and unilateral groups. The predicted difference at the end of treatment was 1.08 (95% confidence interval [CI] = -1.67 to 3.84; p < 0.05, Regression, Linear — Primary statistical analysis was assessment of difference in HAM-D scores between arms at end-of-treatment, supplemented by 95% CIs and this interval compared with the pre-specified noninferiority threshold (-4 points). The p-value was calculated; A regression model was fitted to end-of-treatment HAM-D measures, with baseline HAM-D scores, trial arm, randomization stratifiers as covariates; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [-1.67 to 3.84] — The prespecified noninferiority margin was no more than a -4-point difference at the end of treatment between bitemporal and unilateral groups. The predicted difference at the end of treatment was 1.08 (95% confidence interval [CI]=-1.67 to 3.84)

2. Secondary Outcome: Columbia Autobiographical Memory Interview-Short Form (AMI-SF)
Description: The AMI-SF is used to assess retrospective autobiographical memory function. It has six categories, which involve five questions each, about a family member, most recent travel, last New Year's Eve, last birthday, most recent employment and last visit to a doctor for a physical complaint. At baseline interviewers encourage the participant to recall as much information as they can. Responses at baseline can be scored either two points, for a recognisable real memory, or zero for no memory or too little information to constitute a proper memory. Only those questions for which a memory had been retrieved at baseline are examined at follow-up. Follow-up assessments are scored as percentage recall of baseline score, which is scored as 100% irrespective of actual performance..
Time Frame: end of allocated ECT course
Population: Not all patients completed this cognitive task.
Measure: Mean (Standard Deviation); unit: % of baseline performance
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Number analyzed (Participants) | 64 | 64
% of baseline performance | 56.8 (17.3) | 67.1 (16.3)
Statistical Analysis 1: Comparison: Bilateral ECT Mecta 5000M vs High-dose Unilateral ECT Mecta 5000M; The AMI-SF at end of treatment was analyzed using generalized linear models with a binomial distribution and logit-link. Post treatment AMI-SF measures provide the number of baseline items recalled after ECT; such "number of items recalled" variables were therefore modeled as arising from binomial distributions, with maximum number of possible recalls set to the number of items obtained at baseline; Test type: Superiority or Other; p = 0.001, generalized linear models with a binomia — As above; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.51 to 0.85]

3. Secondary Outcome: Columbia Autobiographical Memory Interview-Short Form (AMI-SF)
Description: as for outcome 2
Time Frame: 3 months follow-up
Population: Not all patients completed this cognitive task.
Measure: Mean (Standard Deviation); unit: % of baseline performance
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Number analyzed (Participants) | 48 | 56
% of baseline performance | 56.2 (18.1) | 67.3 (14.2)
Statistical Analysis 1: Comparison: Bilateral ECT Mecta 5000M vs High-dose Unilateral ECT Mecta 5000M; Test type: Superiority; p = 0.001, Regression, Linear; Analyzed using a generalized linear models with a binomial distribution and logit-link; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.45 to 0.78]

4. Secondary Outcome: Columbia Autobiographical Memory Interview-Short Form (AMI-SF)
Description: as for outcome 2
Time Frame: 6 months follow-up
Population: Not all patients completed this cognitive task.
Measure: Mean (Standard Deviation); unit: % of baseline performance
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Number analyzed (Participants) | 42 | 49
% of baseline performance | 52.9 (16.4) | 63.4 (17.7)
Statistical Analysis 1: Comparison: Bilateral ECT Mecta 5000M vs High-dose Unilateral ECT Mecta 5000M; Test type: Superiority; p = 0.001, Regression, Linear; generalized linear models with a binomial distribution and logit-link; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.45 to 0.79]

ADVERSE EVENTS:
Time Frame: Participants were monitored for ECT-related adverse events during individual ECT sessions and throughout the ECT treatment course, an average of four weeks per participant. They were also monitored for any other adverse events (not directly related to treatment with ECT) throughout the six month follow-up.
Arm/Group | Bilateral ECT Mecta 5000M | High-dose Unilateral ECT Mecta 5000M
Serious Adverse Events (participants affected / at risk) | 9/69 | 7/69
Other Adverse Events (participants affected / at risk) | 33/69 | 37/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral ECT Mecta 5000M (N=69) | High-dose Unilateral ECT Mecta 5000M (N=69)
ECT-related hypertension (Cardiac disorders) | 2 (2) | 4 (4) — required beta-blockers for ECT-related hypertension
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — one patient developed laryngospasm with temporary drop in oxygen saturation
tachyarrhythmia (Cardiac disorders) | 1 (1) | 1 (1) — one patient developed tachyarrhythmia necessitating ECT termination
attempted suicide (Psychiatric disorders) | 0 (0) | 1 (1) — one patient attempted suicide during the course of ECT
interictal confusion (Nervous system disorders) | 3 (3) | 0 (0) — three patients developed interictal confusion resulting in postponement/termination of ECT
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — one patient developed a pulmonary embolus after the fifth treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral ECT Mecta 5000M (N=69) | High-dose Unilateral ECT Mecta 5000M (N=69)
Headache (Nervous system disorders) | 19 (19) | 18 (18) — Post ECT headache, mild and transient
nausea (Gastrointestinal disorders) | 8 (8) | 11 (11) — post ECT nausea, requiring anti emetic
muscle pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) — post ECT muscle pain, mild and transient

LIMITATIONS AND CAVEATS:
We did not include involuntary patients who could not consent due to illness severity (7.4% of referrals), for whom bitemporal ECT may be better. The AMI-SF does not allow quantification of retrograde amnesia attributable directly to ECT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes